CLINICAL TRIAL: NCT00550342
Title: Anti-CD20, Rituximab, for the Treatment of Recurrent or Primary Resistant Focal Segmental Glomerulosclerosis (FSGS)
Brief Title: Rituximab Treatment of Focal Segmental Glomerulosclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Problems with drug supply
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Genentech, Inc. (Industry); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21 DK77329 (completed); R21DK077329 (NIH)
Record Dates: First submitted 2007-10-26; First posted 2007-10-29 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2012-04

CONDITIONS: Focal Segmental Glomerulosclerosis (FSGS)
Keywords: Focal segmental glomerulosclerosis; FSGS; Proteinuria; rituximab; B cell; autoimmune; CD20; treatment; children
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Proteinuria | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab (Experimental): Rituximab (375 mg/m2) will be administered intravenously as per current package label in a facility capable of handling infusion reactions. Subjects would be pre dosed with diphenhydramine and acetaminophen. Solu-Medrol, 1.5 mg/kg would be dosed 1 hour prior to the first dose of rituximab. Three subsequent doses of rituximab will be given at weekly intervals.
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — 375 mg/m2 intravenously for 4 doses
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to determine whether the approved drug, rituximab, is effective in the treatment of focal segmental glomerulosclerosis (FSGS)

DETAILED DESCRIPTION:
Focal segmental glomerulosclerosis (FSGS) remains an enigmatic disease despite many years of study. There has been a recent increased incidence of FSGS particularly in African Americans in whom the outcome tends to be worse. In about 30% of patients transplanted for FSGS, the disease recurs and often results in severe nephrotic syndrome and accelerated graft loss. FSGS is a common cause of nephrotic disease accounting for 10-20% of cases of idiopathic nephrotic syndrome in children and 35% of cases in adults. Most cases are refractory to current therapy resulting in the ultimate progression to end stage renal disease. Overall, FSGS accounts for about 15% of pediatric and 5% of adult cases of end stage renal disease. With the frequent post transplant recurrence, the morbidity and mortality of FSGS is increased. Thus, FSGS is a disease that is associated with a large cost to society and long-term morbidity to the individual patient. A treatment that could induce permanent remission and reverse organ damage would make a major contribution to society by reduction of these expenses. A circulating Permeability Factor (PF, Savin Factor) has been suspected as central to the pathogenesis of recurrent disease but its identity has been difficult to discern. The molecular weight has reported to be between 30 and 100 kDa. Although, PF has been reported to adhere to protein A columns and such columns can be part of the treatment of FSGS, this molecular weight would exclude PF being an intact antibody. Immunosuppressive agents have been the only therapy demonstrating efficacy, albeit partial, suggesting that at least some cases of FSGS are immune mediated. While high dose steroids are the first line of treatment for FSGS, cyclosporine has been efficacious in randomized trials and has been used for steroid resistant FSGS but is associated with substantial toxicity. If cyclosporine fails, cyclophosphamide, plasmapheresis, protein A immunoabsorption, and most recently mycophenolate mofetil (MMF) have been used with variable efficacy.

Rituximab, primarily indicated for treatment of lymphoma, has become a first line agent in the treatment of post transplant lymphoma. However, it has been used with increased frequency to treat various autoimmune diseases including those such as rheumatoid arthritis that have been thought to be primarily T-cell mediated and others such as immune thrombocytopenia purpura that have been thought to be primarily B-cell mediated. In a trial being conducted by the Immune Tolerance Network, ANCA positive vasculitis is being treated with rituximab and it appears that a short course of rituximab leads to tolerance in this autoimmune disease. Rituximab's mechanism of action in the various autoimmune diseases for which has efficacy has been variously suggested to result from elimination of either circulating autoantibody, by elimination of B-cell produced cytokines, or by interference with the antigen presentation provide by B cells.

We have recently had a case of immediate post transplant recurrence of FSGS in a child that failed to respond to MMF, steroids, long-term plasmapheresis and conversion from tacrolimus to cyclosporine. The FSGS associated proteinuria however completely resolved at about 6 months after treatment of post transplant lymphoma with 6 doses of rituximab. A similar case that also resolved after treatment of PTLD with rituximab was recently reported. While the mechanism of action of both cyclosporine and MMF is unknown in FSGS, both drugs have been shown to have activity against B cells. The response seen in these two recent cases following treatment with a B cell specific agent leads to the hypothesis that at least some cases of FSGS have an autoimmune mechanism in which B cells play a central role. We propose to test this hypothesis by the treatment of patients with recurrent or primary persistent FSGS with rituximab.

This study will be a single center, single-arm, pilot trial. As the study will be registered at clintrials.gov, subjects may be referred from outside physicians. However, all treatment will be done at IU in the GCRC. After meeting inclusion/exclusion criteria and signing the consent, serum for PF levels, and blood for B cell flow cytometry will be obtained. Rituximab (375 mg/m2) will be administered intravenously as per current package label in a facility capable of handling infusion reactions. Subjects would be pre dosed with diphenhydramine and acetaminophen. Solu-Medrol, 1.5 mg/kg would be dosed 1 hour prior to the first dose of rituximab. Three subsequent doses of rituximab will be given at weekly intervals. Study visits will then be conducted monthly thereafter for the 6 months and then every 3 months, at which time, assessments of safety will be made. Efficacy will be determined by monitoring first AM Uprotein/C ratio. Flow cytometry, PF factor, urine proteomics and general blood work including CBC, Chemistry, electrolytes, serum immunoglobulin will also be done. During the second year, subjects would be followed every three months. The primary endpoint will be resolution of proteinuria defined as a Up/C ratio of <0.2. Secondary endpoints will be the number of subjects who achieve partial remission defined at a fall of 50% or more in the Up/C ratio from the pre-treatment baseline; the number of patients who develop a recurrence or increase of proteinuria on samples obtained at least 4 weeks apart; effect of treatment on PF levels; safety as measured by infections and drug infusion reactions. Consideration will be given to a plan of redosing in subjects who relapse after initial response.

ELIGIBILITY:
Inclusion Criteria:

1. Primary FSGS involving either native kidneys or primary FSGS recurring after renal transplantation. Age 5-60 years at onset of signs or symptoms of FSGS
2. Estimated GFR ≥ 40 ml/min/1.73 m2
3. Up/c > 1.0 g protein/g creatinine on first am void
4. Biopsy confirmed as primary FSGS (including all subtypes). At least 1 glomerulus demonstrating segmental sclerosis or minimal change FSGS or idiopathic mesangial proliferation with negative immunostains by light microscopy and no dense deposits on electron microscopy. Biopsy required but can be normal for those subjects with rapid recurrence of post transplant FSGS.
5. Steroid resistance as defined by primary physician
6. If participant is female with reproductive potential, she must be willing to avoid pregnancy and have a negative pregnancy test
7. At least one month from last immunization received

Exclusion Criteria:

1. Are immunodeficient or have clinically significant chronic lymphopenia
2. Have an active infection or positive PPD test result
3. Be currently pregnant or lactating, or anticipate getting pregnant
4. Have serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C infection
5. Have any complicating medical issues that interfere with study conduct or cause increased risk
6. Have a history of malignancies within the last five years except for adequately treated skin cancer
7. Have severe cardiac problems such as angina or medically treated arrythmia

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be resolution of proteinuria defined as a Up/C ratio of <0.2. | One year

SECONDARY OUTCOMES:
Number of subjects who achieve partial remission defined at a fall of 50% or more in the Up/C ratio from the pre-treatment baseline | one year
Number of subjects who develop a recurrence or increase of proteinuria on samples obtained at least 4 weeks apart | one year
Effect of treatment on PF levels | one year
Safety as measured by infections and drug infusion reactions. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Pescovitz, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Pescovitz MD, Book BK, Sidner RA. Resolution of recurrent focal segmental glomerulosclerosis proteinuria after rituximab treatment. N Engl J Med. 2006 May 4;354(18):1961-3. doi: 10.1056/NEJMc055495. No abstract available. PMID 16672715